CLINICAL TRIAL: NCT07024862
Title: Long-Term Real-World Outcomes Among Patients With Programmed Death-Ligand 1 (PD-L1) <1% Metastatic Non-Small Cell Lung Cancer (mNSCLC) Treated With First-Line (1l) Nivolumab + Ipilimumab + 2 Cycles Of Chemotherapy (NIC)
Brief Title: Long-term Outcomes Among Patients With Programmed Death-ligand 1 <1% Metastatic Non-small Cell Lung Cancer Treated With First-line Nivolumab + Ipilimumab + 2 Cycles of Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1496
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: Metastatic non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Adults diagnosed with programmed death-ligand 1 (PD-L1) <1% metastatic non-small cell lung cancer (mNSCLC) treated with first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy (NIC) in the US
  Interventions: Biological: nivolumab + ipilimumab

INTERVENTIONS:
Biological: nivolumab + ipilimumab — First-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy (NIC)

SUMMARY:
The study will assess the long-term real-world outcomes among adults diagnosed with programmed death-ligand 1 (PD-L1) <1% metastatic non-small cell lung cancer (mNSCLC) treated with first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy (NIC) in the US

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at confirmed diagnosis with metastatic non-small cell lung cancer (NSCLC) (stage IV), squamous or non-squamous histology
* Initiated first-line (1L) combination nivolumab, ipilimumab, and 2 cycles of platinum-doublet chemotherapy (NIC) regimen between 01 January 2018 and 2 years prior to study launch
* Tumor programmed death-ligand 1 (PD-L1) negative expression (i.e., PD-L1 <1%)
* No EGFR, ALK, or ROS1 genetic mutation (i.e., wild type)
* Minimum of 6 months of follow-up after initiation of 1L NIC*

Exclusion Criteria:

• Any prior systemic therapy for metastatic non-small cell lung cancer (NSCLC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults diagnosed with programmed death-ligand 1 (PD-L1) <1% metastatic non-small cell lung cancer (NSCLC) and treated with 1L combination nivolumab, ipilimumab, and 2 cycles of platinum-doublet chemotherapy (NIC) in the US community oncology setting
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant baseline socio-demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant treatment history | Baseline
Treatment start and stop dates | Up to 6-months
Reasons for 1L treatment selection | Day 1
Initial 1L NIC treatment dose received | Day 1
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Type of chemotherapy received as part of NIC treatment | Day 1
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Participant NIC treatment chemotherapy schedule | Day 1
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Number of NIC treatment interruptions | Up to 6-months
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Date(s) of NIC treatment interruptions | Up to 6-months
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Reasons for NIC treatment interruptions | Up to 6-months
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Length of NIC treatment delay/interruption | Up to 6-months
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Reasons for NIC treatment discontinuation | Up to 6-months
  NIC = first-line (1L) nivolumab + ipilimumab + 2 cycles of chemotherapy
Type of 2L treatment received | Up to 6-months
Reasons for not initiating 2L treatment | Up to 6-months
Start and stop dates of 2L treatment initiation | Up to 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cardinal Health, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts